CLINICAL TRIAL: NCT05265533
Title: Measurement of Body Weight Using Smart Shoe Insole Pressure Sensors
Brief Title: Measurement of Body Weight Using Shoe Insole Pressure Sensors
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Susan Roberts, Senior Scientist, Tufts University
Other Study IDs: STUDY00001324
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Effect of Different Weights

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to create a dataset to help accelerate machine learning (ML) based solutions for applications such as activity recognition, detect changes in weight and predict weight of carried load. The research will further help in the development of novel machine learning-based algorithm for accurately predicting the body weight of an individual in real-time and within few ounces error margin, using sampled data from smart insole sensors.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 18-70 years

Exclusion Criteria:

* Refusal to adhere to covid19 safety guidelines

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Convenient sample recruited within Tufts University
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Pressure readings | 1hr

CONTACTS AND LOCATIONS:
Locations (1):
- Susan Roberts, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan on sharing the de-identified data collected with other researchers